CLINICAL TRIAL: NCT03940183
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Trelagliptin Succinate Monotherapy for Type 2 Diabetes
Brief Title: Clinical Trial of Trelagliptin Succinate Tablets in the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC/HC1425/201801
Record Dates: First submitted 2019-04-15; First posted 2019-05-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; monotherapy; trelagliptin succinate
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trelagliptin succinate 100 mg (Experimental): Tablets,100mg per tablet,oral, once a week, 100mg each time, continuous medication for a total of 24 weeks
  Interventions: Drug: Trelagliptin Succinate
- Placebo Oral Tablet (Placebo Comparator): Tablets,N/A,oral, once a week, one tablet each time, continuous medication for a total of 24 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Trelagliptin Succinate — the experimental group will use trelagliptin succinate 100 mg for 24weeks
  Arms: Trelagliptin succinate 100 mg
Drug: Placebo Oral Tablet — the placebo Comparator groups use placebo oral tablet for 24weeks
  Arms: Placebo Oral Tablet

SUMMARY:
The trial used a randomized, double-blind, placebo-controlled, superior-effect design, multicenter clinical study.

The trial was divided into a test group and a placebo group,the two groups were randomized in a 1:1 ratio and planned to enroll 240 patients with type 2 diabetes. After 2 weeks of screening, all subjects entered the treatment period,which was 24 weeks, and 1 week period of follow-up.

DETAILED DESCRIPTION:
The trial was divided into a test group and a placebo group: the test group was given trelagliptin succinate tablets, and the placebo group was given placebo. The test group and the placebo group were randomized in a 1:1 ratio and planned to enroll 240 patients with type 2 diabetes. After 2 weeks of screening, all subjects entered the treatment period,which was 24 weeks, and 1 week period of follow-up.

All subjects were asked to continue their current diabetes diet and physical activity treatment plan throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who fully understand the test content and possible adverse reactions and voluntarily participate in the trial and sign the informed consent form;
* Subjects who meet the World Health Organization(WHO) (1999) criteria for the diagnosis and classification criteria for type 2 diabetes;
* 18 ≤ age ≤ 75 years old, male or female;
* One of the following conditions:

  * Initially diagnosed type 2 diabetic patients;
  * Patients who with type 2 diabetes diagnosed within 2 years of screening period and are treated with single-agent oral hypoglycemic agents until screening, and do not take the medicine regularly for at least 8 weeks (ie, continuous medication for <1 week);
* 19kg/m^2 ≤ Body Mass Index（BMI ）≤ 35kg/m^2;
* 7.0% ≤ HbA1c ≤ 10.0%;
* Female subjects of childbearing age are negative in pregnancy test;
* Female subjects do not have a fertility plan one month before the trial and all the subjects do not have a fertility plan during and one month after the trial.

Exclusion Criteria:

* Fasting plasma glucose≥13.9mmol/L or a history of severe hypoglycemia (blood sugar below 2.8mmol/L);
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg during screening;
* Positive for Acquired Immure Deficiency Syndrome（AIDS）or syphilis testing;
* Active hepatitis B virus infection or hepatitis C virus infection;
* History of acute or chronic liver disease, and Aspartate aminotransferase(AST) or Alanine minotransferase(ALT)> 2.5 times of reference range or total bilirubin> 1.5 times of reference range during the screening period;
* Renal insufficiency subjects, the serum creatinine above 1.5 times of reference range during the screening period;
* The white blood cells are outside of the reference range, hemoglobin below the reference range, triglyceride>5.7mmol/L during the screening period;
* Acute complications of diabetes (including diabetic ketoacidosis, hyperosmolar nonketotic diabetic coma, lactic acidosis and hypoglycemia coma) ,or severe chronic complications (proliferative diabetic retinopathy, diabetic nephropathy);
* Oral or intravenous use of glucocorticoids or regular application (ie continuous use more than one week within 4 weeks before screening time) with large doses of thiazide diuretics (hydrochlorothiazide, chlorothiazide, etc.);
* Subjects without a pacemaker, the 12-lead ECG showed II or III degree atrioventricular block, long QT syndrome or corrected QT interval （QTc）>450ms or atrial fibrillation during the screening period;
* Active heart disease (including acute myocardial infarction, unstable angina) , moderate to severe congestive heart failure (NYHA class III or IV), or planned for coronary artery bypass grafting or transmyocardial laser revascularization half year before the screening period.
* History of epilepsy, mental illness, major depression,or previous thyroid function abnormal and still being treated, or those with organ transplants, severe chronic lung disease, and other serious heart disease, cerebrovascular disease, blood disease;
* Endocrine diseases such as hypercortisolism or polycystic ovary syndrome that may affect blood glucose levels;
* Inflammatory bowel disease, colon ulcer, partial intestinal obstruction or obvious digestive and dysfunction chronic bowel disease;
* Active pancreatitis, cholecystitis, gallstones and other digestive diseases;
* Using weight loss surgery within 3 months before screening period or using weight-loss drugs (including traditional Chinese medicine diet pills) within2 months before screening period;
* History of drug or drug abuse or alcoholics;
* Blood donation within 2 months before screening includes blood components or massive blood loss (≥400mL),or receiving blood transfusion or using blood products;
* History of allergies with similar drugs (DPP-4 inhibitors) or those who are judged by the investigator to be allergic to the test drug;
* Subjects who are participating in other clinical trials or who have participated in other drug trials within 3 months prior to screening;
* Pregnancy (defined as positive in pregnancy test), lactating women;
* Not suitable for this clinical trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, week 24
  Changes in HbA1c compared to baseline at week 24

SECONDARY OUTCOMES:
HbA1c | Baseline, week 16
  Changes in HbA1c compared to baseline at week 16
Fasting blood glucose | Baseline, week 16，week 24
  Changes in Fasting blood glucose compared to baseline at week 16,week 24
2-hour postprandial blood glucose | Baseline, week 24
  Changes in 2-hour postprandial blood glucose compared to baseline at week 24
fasting insulin | Baseline, week 24
  Changes in fasting insulin compared to baseline at week 24
fasting glucagon | Baseline, week 24
  Changes in fasting glucagon compared to baseline at week 24
active Glucagon-like peptide-1（GLP-1） level | Baseline, week 24
  Changes in active Glucagon-like peptide-1（GLP-1） level compared to baseline at 24
The percentage of HbA1c<6.5% and HbA1c<7% | week 24
  The percentage of HbA1c<6.5% and HbA1c<7% at week 24
body weight | Baseline, week 24
  Changes in body weight（Kg）compared to baseline at week 24
Body Mass Index | Baseline, week 24
  Changes in Body Mass Index （kg/m^2）compared to baseline at week 24

CONTACTS AND LOCATIONS:
Overall Officials: yueying peng, Study Chair — Clinical Medicine Department CSPC R&D Business Division
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No